CLINICAL TRIAL: NCT03572062
Title: A PHASE 1/2, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLIND,DOSE-FINDING, FIRST-IN-HUMAN STUDY TO DESCRIBE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF AN ADJUVANTED RESPIRATORY SYNCYTIAL VIRUS (RSV) VACCINE IN HEALTHY OLDER ADULTS
Brief Title: A Study to Evaluate the Safety and Immunogenicity of an Adjuvanted RSV Vaccine in Healthy Older Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely by sponsor and will not resume, participants are no longer being examined or receiving intervention.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671002; RSV ADJUVANT (Other: Alias Study Number)
Record Dates: First submitted 2018-06-01; First posted 2018-06-28 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Tract Infection
Keywords: Respiratory tract infection, RSV, Adjuvant, vaccine
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Arm 1 (Experimental): Low dose formulation A and SIIV
  Interventions: Biological: Formulation A
- Arm 2 (Experimental): Low dose formulation B and SIIV
  Interventions: Biological: Formulation B
- Arm 3 (Experimental): Mid dose formulation A and SIIV
  Interventions: Biological: Formulation A
- Arm 4 (Experimental): Mid dose formulation B and SIIV
  Interventions: Biological: Formulation B
- Arm 5 (Experimental): High dose formulation A and SIIV
  Interventions: Biological: Formulation A
- Arm 6 (Experimental): High dose formulation B and SIIV
  Interventions: Biological: Formulation B
- Arm 7 (Experimental): High dose formulation C and SIIV
  Interventions: Biological: Formulation C
- Arm 8 (Placebo Comparator): Placebo and SIIV
  Interventions: Biological: Placebo
- M0M2 Arm 1 (Experimental): High dose formulation B
  Interventions: Biological: Formulation B
- M0M2 Arm 2 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Formulation A — RSV vaccine
  Arms: Arm 1; Arm 3; Arm 5
Biological: Formulation B — Adjuvanted RSV vaccine
  Arms: Arm 2; Arm 4; Arm 6; M0M2 Arm 1
Biological: Formulation C — RSV vaccine
  Arms: Arm 7
Biological: Placebo — Placebo
  Arms: Arm 8; M0M2 Arm 2

SUMMARY:
The study will evaluate the safety, tolerability, and immunogenicity of up to 7 different RSV vaccine candidates, some with adjuvant, when administered concomitantly with seasonal inactivated influenza vaccine (SIIV) and may evaluate a second dose of RSV vaccine administered12 months after the initial dose.

In addition the study will evaluate a 2-dose regimen administered 2 months apart to 62 subjects.

DETAILED DESCRIPTION:
The study will evaluate the safety, tolerability, and immunogenicity of up to 7 different RSV vaccine candidates, some with adjuvant, when administered concomitantly with SIIV. Healthy male and female subjects between 65 to 85 years of age will be enrolled. Subjects will receive 2 intramuscular injections to assess the concomitant administration of SIIV when given to subjects receiving one of the 3 RSV vaccine dose-level candidates formulated with or without an adjuvant.

If interim support implementation of revaccination, invited, consenting subjects will be revaccinated with the same dose and formulation of the RSV vaccine or placebo received at Visit 1, concomitantly with SIIV. The safety, tolerability, and immunogenicity of the second dose will be evaluated through 12 months after revaccination.

62 subjects will be randomized 1:1 to receive a dose of high dose adjuvanted RSV vaccine or placebo followed by a second dose 2 months later. Safety, tolerability, and immunogenicity will be evaluated. The subjects will be enrolled before the influenza season. There will be no concomitant SIIV administration.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject has been informed of all pertinent aspects of the study.
2. Healthy adults who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
3. Willing and able to comply with scheduled visits, vaccination plan, laboratory tests, and other study procedures.
4. Male and nonchildbearing-potential female adults aged 65 to 85 years at the time of enrollment (signing of the ICD).
5. Subjects must have received the primary vaccination (RSV vaccine or placebo) at Visit 1 and have signed and dated the ICD for participating in the revaccination stage (applies to Primary Study Cohort - Stage 2 subjects).

Exclusion Criteria:

1. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
2. Participation in other studies involving investigational product within 28 days prior to study entry and/or during study participation.
3. Known infection with HIV, hepatitis C virus (HCV), or hepatitis B virus (HBV).
4. Previous vaccination with any licensed or investigational RSV vaccine before enrollment into the study, or planned receipt throughout the study of nonstudy RSV vaccine.
5. Vaccination with any influenza vaccine within 6 months (182 days) before investigational product administration (applies to Primary Study Cohort - Stages 1 and 2).
6. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the investigational product(s), including natural rubber latex. In addition, a history of severe allergic reaction (eg, anaphylaxis) to any substance, including documented allergy to egg proteins (egg or egg products) or chicken proteins.
7. Subjects with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
8. Subjects who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, subjects should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before investigational product administration.Inhaled/nebulized, intra-articular, intrabursal, or topical (epidural, skin or eyes) corticosteroids are permitted.
9. Subject with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention including but not limited to: systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome,multiple sclerosis, Sjögren syndrome, idiopathic thrombocytopenic purpura, autoimmune glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and insulin-dependent diabetes mellitus (type 1).
10. Receipt of blood/plasma products or immunoglobulin, from 60 days before investigational product administration or planned receipt throughout the study.
11. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
12. Female subjects of childbearing potential or who are pregnant or breastfeeding; fertile male subjects who are unwilling to use a highly effective method of contraception for at least 28 days after the last dose of investigational product.
13. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
14. Planned donation of blood volumes of approximately 470 mL within 12 weeks after Vaccination 1 (applies to subjects having additional blood drawn for cellular assays).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 317 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (4):
  - Qps Mra, Llc, South Miami, Florida
  - Optimal Research, LLC, Peoria, Illinois
  - Synexus Clinical Research US, Fremont, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
- Australia (12):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - AIM Centre (Hunter Diabetes Centre), Merewether, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Westmead Hospital (Infectious Diseases and Microbiology), Westmead, New South Wales
  - Data Health Australia Pty Limited (Trading as AusTrials), Taringa, Queensland
  - Eastern Health, Box Hill, Victoria
  - Emeritus Research Pty. Ltd., Camberwell, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Barwon Health, Geelong, Victoria
  - Doctors of Ivanhoe, Ivanhoe, Victoria
  - Institute for Respiratory Health, Nedlands, Western Australia
  - TrialsWest, Spearwood, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Baber J, Arya M, Moodley Y, Jaques A, Jiang Q, Swanson KA, Cooper D, Maddur MS, Loschko J, Gurtman A, Jansen KU, Gruber WC, Dormitzer PR, Schmoele-Thoma B. A Phase 1/2 Study of a Respiratory Syncytial Virus Prefusion F Vaccine With and Without Adjuvant in Healthy Older Adults. J Infect Dis. 2022 Dec 13;226(12):2054-2063. doi: 10.1093/infdis/jiac189. PMID 35543281
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in 2 Cohorts: Primary Cohort (Single administration of RSVpreF formulations or placebo, co-administered with seasonal inactivated influenza vaccine [SIIV]), and Month-0, Month-2 Cohort (two doses of an RSVpreF formulation or placebo administered two months apart).
Groups:
- Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV: Participants were administered an intramuscular dose of respiratory syncytial virus stabilized prefusion F subunit (RSVpreF) 60 microgram (mcg) with aluminum hydroxide (Al[OH]3) by injecting 0.5 milliliter (mL) dose along with single 0.5mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV: Participants were administered an intramuscular dose of RSVpreF 60 mcg with CpG/Al(OH)3 as 0.5-mL injection along with single 0.5 mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV: Participants were administered an intramuscular dose of RSVpreF 120 mcg with Al(OH)3 as 0.5-mL injection along with single 0.5 mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV: Participants were administered an intramuscular dose of RSVpreF 120 mcg with CpG/Al(OH)3 as 0.5-mL injection along with single 0.5 mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV: Participants were administered an intramuscular dose of RSVpreF 240 mcg with Al(OH)3 as 0.5-mL injection along with single 0.5 mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV: Participants were administered an intramuscular dose of RSVpreF 240 mcg with CpG/Al(OH)3 as 0.5-mL injection along with single 0.5 mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Primary Cohort: RSVpreF 240 mcg + SIIV: Participants were administered an intramuscular dose of RSVpreF 240 mcg as 0.5-mL injection along with single 0.5 mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Primary Cohort: Placebo + SIIV: Participants were administered an intramuscular dose of placebo intramuscularly as 0.5-mL injection along with single 0.5 mL intramuscular dose of SIIV on Day 1. Participants were followed-up through Month 12.
- Month-0, Month-2 Cohort: RSVpreF 240 mcg + CpG/Al(OH)3: Participants were administered an intramuscular dose of RSVpreF 240 mcg with CpG/Al(OH)3 as 0.5-mL injection on Day 1 Month 0 (Vaccination 1) and Month 2 (Vaccination 2: 54 to 66 Days after Vaccination 1). Participants were followed up through 6 months after Vaccination 2.
- Month-0, Month-2 Cohort: Placebo: Participants were administered an intramuscular dose of placebo as 0.5-mL injection on Day 1 Month 0 (Vaccination 1) and Month 2 (Vaccination 2: 54 to 66 Days after Vaccination 1). Participants were followed up through 6 months after Vaccination 2.
Period: Overall Study
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV | Month-0, Month-2 Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 | Month-0, Month-2 Cohort: Placebo
Started | 32 | 32 | 32 | 31 | 32 | 32 | 32 | 31 | 32 | 31
Treated | 32 | 32 | 32 | 31 | 31 | 30 | 32 | 30 | 32 | 31
Completed | 32 | 32 | 32 | 31 | 31 | 28 | 31 | 30 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 32 | 31
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 27
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Randomized But Not Treated | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of the investigational products (RSVpreF or placebo) at Visit 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV | Month-0, Month-2 Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 | Month-0, Month-2 Cohort: Placebo | Total
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 31 | 30 | 32 | 30 | 32 | 31 | 313
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean | 71.2 (5.4) | 71.0 (4.8) | 72.3 (4.5) | 70.2 (4.3) | 71.4 (5.3) | 70.2 (3.5) | 70.4 (5.4) | 70.8 (4.5) | 72.2 (4.4) | 72.6 (5.4) | 71.2 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 17 | 16 | 13 | 11 | 12 | 14 | 16 | 17 | 145
  Male | 15 | 20 | 15 | 15 | 18 | 19 | 20 | 16 | 16 | 14 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 32 | 32 | 32 | 31 | 30 | 30 | 32 | 30 | 32 | 31 | 312
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 2 | 3 | 1 | 1 | 3 | 4 | 4 | 1 | 2 | 23
  Race: White | 30 | 30 | 29 | 29 | 29 | 27 | 26 | 25 | 31 | 29 | 285
  Race: Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Race: Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Primary Cohort: Percentage of Participants With Local Reactions Within 14 Days After Vaccination 1
Description: Local reactions included redness, swelling, and pain at the injection site (left arm) recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units (range: 1 to 20, and greater than [>] 21). 1 measuring device unit = 0.5 centimeter (cm) and graded as: mild (2.5 to 5.0 cm), moderate (greater than [>] 5.0 to 10.0 cm), and severe (>10 cm). Pain at injection site was graded as: mild (did not interfere with activity), moderate (interferes with activity) and severe (prevented daily activity).
Time Frame: Within 14 days after Vaccination 1
Population: Safety population included all participants who received at least 1 dose of the investigational products (RSVpreF or placebo) at Visit 1. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected for Primary cohort only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV
Number analyzed (Participants) | 31 | 32 | 32 | 31 | 31 | 30 | 32 | 30
percentage of participants
  Pain at Injection Site: Mild | 32.3 [16.7 to 51.4] | 28.1 [13.7 to 46.7] | 3.1 [0.1 to 16.2] | 25.8 [11.9 to 44.6] | 22.6 [9.6 to 41.1] | 16.7 [5.6 to 34.7] | 18.8 [7.2 to 36.4] | 6.7 [0.8 to 22.1]
  Pain at Injection Site: Moderate | 0 [0.0 to 11.2] | 3.1 [0.1 to 16.2] | 0 [0.0 to 10.9] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 3.3 [0.1 to 17.2]
  Pain at Injection Site: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Redness: Mild | 3.2 [0.1 to 16.7] | 0 [0.0 to 10.9] | 3.1 [0.1 to 16.2] | 0 [0.0 to 11.2] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 3.1 [0.1 to 16.2] | 0 [0.0 to 11.6]
  Redness: Moderate | 3.2 [0.1 to 16.7] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 3.1 [0.1 to 16.2] | 0 [0.0 to 11.6]
  Redness: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Swelling: Mild | 3.2 [0.1 to 16.7] | 3.1 [0.1 to 16.2] | 3.1 [0.1 to 16.2] | 0 [0.0 to 11.2] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 3.3 [0.1 to 17.2]
  Swelling: Moderate | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Swelling: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]

2. Primary Outcome: Primary Cohort: Percentage of Participants With Systemic Events Within 14 Days After Vaccination 1
Description: Systemic events included fever, fatigue/tiredness, headache, vomiting, nausea, diarrhea, muscle pain and joint pain recorded by participants in an e-diary. Fever was graded as: mild (38.0 to 38.4 degrees [deg] Celsius [C]), moderate (38.5 to 38.9 deg C), severe (39 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle and joint pain were graded as: mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily routine activity). Vomiting was graded as: mild (1-2 times in 24 hours [h]), moderate (>2 times in 24h) and severe (required intravenous hydration). Diarrhea was graded as: mild (2-3 loose stools in 24h), moderate (4-5 loose stools in 24h) and severe (6 or more loose stools in 24h).
Time Frame: Within 14 days after Vaccination 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV
Number analyzed (Participants) | 31 | 32 | 32 | 31 | 31 | 30 | 32 | 30
percentage of participants
  Fever: Mild | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 9.4 [2.0 to 25.0] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Fever: Moderate | 3.2 [0.1 to 16.7] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Fever: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Fever: Grade 4 | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Nausea: Mild | 9.7 [2.0 to 25.8] | 3.1 [0.1 to 16.2] | 3.1 [0.1 to 16.2] | 0 [0.0 to 11.2] | 6.5 [0.8 to 21.4] | 0 [0.0 to 11.6] | 6.3 [0.8 to 20.8] | 10.0 [2.1 to 26.5]
  Nausea: Moderate | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 6.5 [0.8 to 21.4] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Nausea: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Vomiting: Mild | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Vomiting: Moderate | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Vomiting: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 00 [0.0 to 11.6]
  Diarrhea: Mild | 9.7 [2.0 to 25.8] | 3.1 [0.1 to 16.2] | 9.4 [2.0 to 25.0] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2] | 10.0 [2.1 to 26.5] | 6.3 [0.8 to 20.8] | 6.7 [0.8 to 22.1]
  Diarrhea: Moderate | 3.2 [0.1 to 16.7] | 3.1 [0.1 to 16.2] | 6.3 [0.8 to 20.8] | 3.2 [0.1 to 16.7] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 6.7 [0.8 to 22.1]
  Diarrhea: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Headache: Mild | 16.1 [5.5 to 33.7] | 3.1 [0.1 to 16.2] | 3.1 [0.1 to 16.2] | 6.5 [0.8 to 21.4] | 3.2 [0.1 to 16.7] | 16.7 [5.6 to 34.7] | 25.0 [11.5 to 43.4] | 6.7 [0.8 to 22.1]
  Headache: Moderate | 3.2 [0.1 to 16.7] | 6.3 [0.8 to 20.8] | 0 [0.0 to 10.9] | 9.7 [2.0 to 25.8] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 9.4 [2.0 to 25.0] | 0 [0.0 to 11.6]
  Headache: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 3.1 [0.1 to 16.2] | 0 [0.0 to 11.6]
  FatigueTtiredness: Mild | 16.1 [5.5 to 33.7] | 15.6 [5.3 to 32.8] | 9.4 [2.0 to 25.0] | 3.2 [0.1 to 16.7] | 16.1 [5.5 to 33.7] | 3.3 [0.1 to 17.2] | 31.3 [16.1 to 50.0] | 16.7 [5.6 to 34.7]
  Fatigue/Tiredness: Moderate | 6.5 [0.8 to 21.4] | 3.1 [0.1 to 16.2] | 18.8 [7.2 to 36.4] | 25.8 [11.9 to 44.6] | 3.2 [0.1 to 16.7] | 10.0 [2.1 to 26.5] | 9.4 [2.0 to 25.0] | 3.3 [0.1 to 17.2]
  Fatigue/Tiredness: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 3.1 [0.1 to 16.2] | 0 [0.0 to 11.6]
  Muscle Pain: Mild | 9.7 [2.0 to 25.8] | 6.3 [0.8 to 20.8] | 6.3 [0.8 to 20.8] | 9.7 [2.0 to 25.8] | 12.9 [3.6 to 29.8] | 10.0 [2.1 to 26.5] | 12.5 [3.5 to 29.0] | 16.7 [5.6 to 34.7]
  Muscle Pain: Moderate | 0 [0.0 to 11.2] | 3.1 [0.1 to 16.2] | 3.1 [0.1 to 16.2] | 3.2 [0.1 to 16.7] | 3.2 [0.1 to 16.7] | 6.7 [0.8 to 22.1] | 6.3 [0.8 to 20.8] | 3.3 [0.1 to 17.2]
  Muscle Pain: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]
  Joint Pain: Mild | 3.2 [0.1 to 16.7] | 0 [0.0 to 10.9] | 6.3 [0.8 to 20.8] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2] | 6.7 [0.8 to 22.1] | 9.4 [2.0 to 25.0] | 10.0 [2.1 to 26.5]
  Joint Pain: Moderate | 0 [0.0 to 11.2] | 3.1 [0.1 to 16.2] | 9.4 [2.0 to 25.0] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 3.3 [0.1 to 17.2]
  Joint Pain: Severe | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6]

3. Primary Outcome: Primary Cohort: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination 1
Description: An AE is any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. AEs included both serious and non-serious adverse events.
Time Frame: Within 1 month after Vaccination 1
Population: Safety population included all participants who received at least 1 dose of the investigational products (RSVpreF or placebo) at Visit 1. Data for this outcome measure was planned to be collected for Primary cohort only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 31 | 30 | 32 | 30
percentage of participants | 21.9 [9.3 to 40.0] | 21.9 [9.3 to 40.0] | 34.4 [18.6 to 53.2] | 29.0 [14.2 to 48.0] | 25.8 [11.9 to 44.6] | 23.3 [9.9 to 42.3] | 21.9 [9.3 to 40.0] | 16.7 [5.6 to 34.7]

4. Primary Outcome: Primary Cohort: Percentage of Participants With Medically Attended Adverse Events (MAEs) and Serious Adverse Events (SAEs) Through 12 Months After Vaccination 1
Description: An MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility. A SAE is any untoward medical occurrence at any dose: results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect.
Time Frame: Up to 12 months after Vaccination 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 31 | 30 | 32 | 30
percentage of participants
  MAEs | 46.9 [29.1 to 65.3] | 59.4 [40.6 to 76.3] | 46.9 [29.1 to 65.3] | 51.6 [33.1 to 69.8] | 54.8 [36.0 to 72.7] | 60.0 [40.6 to 77.3] | 50.0 [31.9 to 68.1] | 50.0 [31.3 to 68.7]
  SAEs | 6.3 [0.8 to 20.8] | 12.5 [3.5 to 29.0] | 12.5 [3.5 to 29.0] | 12.9 [3.6 to 29.8] | 16.1 [5.5 to 33.7] | 13.3 [3.8 to 30.7] | 12.5 [3.5 to 29.0] | 10.0 [2.1 to 26.5]

5. Secondary Outcome: Primary Cohort: Geometric Mean Titers (GMT) of Respiratory Syncytial Virus Subgroup A (RSV A) and Respiratory Syncytial Virus Subgroup B (RSV B) Neutralizing Antibodies Before and 1 Month After Vaccination 1
Description: GMTs of RSV A and RSV B antigens were measured using neutralizing assay. Titers above the lower limit of quantitation (LLOQ) were considered accurate and their quantitated values were reported. The neutralizing titer LLOQ values were: A = 50 and B = 70. Assay results below the LLOQ were set to 0.5 × LLOQ.
Time Frame: Before vaccination and 1 Month after Vaccination 1
Population: Evaluable immunogenicity population: eligible participants who received both SIIV and RSV vaccinations or SIIV and placebo as randomized, had blood drawn within 27-42 days after Visit 1 pre-specified time frames at 1-month post-vaccination follow-up visit, had at least 1 valid, determinate assay result for proposed analysis, had no major protocol violations. Number Analyzed= participants evaluable for each row. Data for this outcome measure was planned to be collected for Primary cohort only.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV
Number analyzed (Participants) | 29 | 32 | 32 | 31 | 31 | 29 | 31 | 30
titers
  RSV A: Before Vaccination 1: number analyzed (Participants) | 29 | 31 | 32 | 31 | 31 | 29 | 31 | 30
  RSV A: Before Vaccination 1 | 2113 [1610.6 to 2772.5] | 2592 [1932.3 to 3477.8] | 2234 [1591.1 to 3136.5] | 2395 [1817.9 to 3155.4] | 2333 [1779.8 to 3057.1] | 2061 [1600.2 to 2653.4] | 2243 [1696.4 to 2966.8] | 2093 [1509.0 to 2903.8]
  RSV A: 1 Month After Vaccination 1 | 15158 [10503.8 to 21875.0] | 12385 [9555.6 to 16051.2] | 17806 [12893.3 to 24590.4] | 15492 [11012.7 to 21793.6] | 18045 [12589.5 to 25865.5] | 23929 [18242.8 to 31386.8] | 23833 [17799.2 to 31912.0] | 1823 [1376.5 to 2415.2]
  RSV B: Before Vaccination 1: number analyzed (Participants) | 29 | 31 | 32 | 31 | 31 | 29 | 31 | 30
  RSV B: Before Vaccination 1 | 1786 [1383.3 to 2305.3] | 2116 [1526.7 to 2933.7] | 1728 [1271.9 to 2346.4] | 2021 [1451.8 to 2812.2] | 1884 [1337.0 to 2655.9] | 1844 [1417.5 to 2398.8] | 1580 [1210.9 to 2061.1] | 1677 [1156.2 to 2433.0]
  RSV B: 1 Month After Vaccination 1 | 15182 [9785.1 to 23555.6] | 9694 [7396.8 to 12705.8] | 14436 [10196.9 to 20436.9] | 12781 [8571.0 to 19058.7] | 18205 [12574.4 to 26356.6] | 20777 [15034.9 to 28711.0] | 22249 [15715.7 to 31497.5] | 1617 [1139.6 to 2294.9]

6. Secondary Outcome: Primary Cohort: Hemagglutination Inhibition Assay (HAI) and Neutralizing Antibody Geometric Mean Titers for All Strains Following the Seasonal Inactivated Influenza Vaccine (SIIV) Before and 1 Month After Vaccination 1
Description: The HAI and neutralizing titer LLOQ value for each strain was 1:10. Assay results below the LLOQ were set to 0.5 × LLOQ. The analysis was performed on following strains: H1N1 A/Michigan, H3N2 A/Brisbane, B/Phuket for HAI and H3N2/Brisbane for neutralizing assay.
Time Frame: Before vaccination and 1 Month after Vaccination 1
Population: Evaluable immunogenicity population: participants who received both SIIV and RSV vaccinations or SIIV and placebo as randomized, had blood drawn within 27-42 days after Visit 1 pre-specified time frames at 1-month post-vaccination follow-up visit, had at least 1 valid, determinate assay result for analysis, had no major protocol violations. Number Analyzed = participants evaluable for each specified row. Data for this outcome was planned to be collected for Primary cohort only.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV
Number analyzed (Participants) | 29 | 32 | 32 | 31 | 31 | 29 | 31 | 30
titers
  HAI: H1N1 A/Michigan: Before Vaccination 1: number analyzed (Participants) | 29 | 31 | 32 | 31 | 31 | 29 | 31 | 30
  HAI: H1N1 A/Michigan: Before Vaccination 1 | 47.9 [31.69 to 72.26] | 42.8 [27.81 to 65.78] | 29.5 [19.03 to 45.84] | 35.8 [22.14 to 57.77] | 37.2 [22.99 to 60.19] | 31.9 [18.31 to 55.48] | 38.3 [27.20 to 53.80] | 35.4 [20.37 to 61.60]
  HAI: H1N1 A/Michigan: 1 Month After Vaccination 1 | 121.5 [84.37 to 175.11] | 114.4 [79.95 to 163.60] | 102.1 [69.15 to 150.65] | 141.5 [90.54 to 221.13] | 143.9 [91.81 to 225.51] | 100.4 [74.68 to 134.96] | 118.3 [84.12 to 166.40] | 149.3 [104.93 to 212.40]
  HAI: H3N2 A/Brisbane: Before Vaccination 1: number analyzed (Participants) | 29 | 31 | 32 | 31 | 31 | 29 | 31 | 30
  HAI: H3N2 A/Brisbane: Before Vaccination 1 | 121.6 [67.92 to 217.54] | 143.9 [90.99 to 227.52] | 57.8 [35.11 to 95.19] | 80.9 [53.49 to 122.38] | 102.3 [61.32 to 170.69] | 90.7 [53.21 to 154.57] | 121.7 [87.32 to 169.55] | 76.8 [45.79 to 128.87]
  HAI: H3N2 A/Brisbane: 1 Month After Vaccination 1 | 297.9 [197.30 to 449.64] | 372.4 [221.98 to 624.70] | 238.9 [167.42 to 340.78] | 251.6 [163.84 to 386.49] | 327.2 [208.41 to 513.80] | 258.1 [174.20 to 382.29] | 286.2 [201.75 to 405.87] | 321.8 [221.41 to 467.83]
  HAI: B/Phuket: Before Vaccination 1: number analyzed (Participants) | 29 | 31 | 32 | 31 | 31 | 29 | 31 | 30
  HAI: B/Phuket: Before Vaccination 1 | 8.7 [6.37 to 11.78] | 8.4 [6.68 to 10.59] | 6.6 [5.61 to 7.82] | 7.9 [6.31 to 9.79] | 8.6 [6.57 to 11.25] | 7.3 [5.55 to 9.69] | 9.1 [6.82 to 12.11] | 7.5 [5.74 to 9.77]
  HAI: B/Phuket: 1 Month After Vaccination 1 | 12.3 [8.99 to 16.90] | 11.2 [8.41 to 14.92] | 10.2 [8.03 to 13.00] | 12.2 [8.62 to 17.15] | 14.4 [10.31 to 20.05] | 14.7 [10.21 to 21.30] | 15.5 [10.86 to 22.02] | 15.2 [10.25 to 22.68]
  Neutralizing assay: H3N2/Brisbane: Before Vaccination 1: number analyzed (Participants) | 29 | 31 | 32 | 31 | 31 | 29 | 31 | 30
  Neutralizing assay: H3N2/Brisbane: Before Vaccination 1 | 12.4 [9.06 to 16.97] | 15.5 [11.94 to 20.02] | 10.2 [8.09 to 12.90] | 9.3 [7.76 to 11.27] | 12.4 [9.03 to 16.93] | 10.1 [7.84 to 13.06] | 12.2 [10.16 to 14.71] | 8.7 [6.92 to 10.95]
  Neutralizing assay: H3N2/Brisbane: 1 Month After Vaccination 1 | 27.3 [19.24 to 38.70] | 27.4 [18.43 to 40.66] | 19.1 [14.63 to 25.06] | 21.4 [16.08 to 28.44] | 22.1 [16.11 to 30.36] | 21.2 [16.15 to 27.90] | 21.9 [16.82 to 28.44] | 26.7 [18.74 to 38.00]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events: within 14 days after vaccination Other AEs: within one month after vaccination; SAEs: Day 1 up to 12 Months for Primary Cohort; Day 1 up to 6 Months for Month-0, Month-2 Cohort
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population included all participants who received at least 1 dose of the investigational products (RSVpreF or placebo) at Visit 1.
Arm/Group | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV | Primary Cohort: RSVpreF 240 mcg + SIIV | Primary Cohort: Placebo + SIIV | Month-0, Month-2 Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 | Month-0, Month-2 Cohort: Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/31 | 0/31 | 1/30 | 0/32 | 0/30 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/32 | 4/32 | 4/32 | 4/31 | 5/31 | 4/30 | 4/32 | 3/30 | 6/32 | 5/31
Other Adverse Events (participants affected / at risk) | 17/32 | 17/32 | 21/32 | 21/31 | 17/31 | 12/30 | 25/32 | 14/30 | 28/32 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV (N=32) | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV (N=32) | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV (N=32) | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV (N=31) | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV (N=31) | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV (N=30) | Primary Cohort: RSVpreF 240 mcg + SIIV (N=32) | Primary Cohort: Placebo + SIIV (N=30) | Month-0, Month-2 Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 (N=32) | Month-0, Month-2 Cohort: Placebo (N=31)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site joint infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Morton's neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort: RSVpreF 60 mcg + Al(OH)3 + SIIV (N=32) | Primary Cohort: RSVpreF 60 mcg + CpG/Al(OH)3 + SIIV (N=32) | Primary Cohort: RSVpreF 120 mcg + Al(OH)3 + SIIV (N=32) | Primary Cohort: RSVpreF 120 mcg + CpG/Al(OH)3 + SIIV (N=31) | Primary Cohort: RSVpreF 240 mcg + Al(OH)3 + SIIV (N=31) | Primary Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 + SIIV (N=30) | Primary Cohort: RSVpreF 240 mcg + SIIV (N=32) | Primary Cohort: Placebo + SIIV (N=30) | Month-0, Month-2 Cohort: RSVpreF 240 mcg + CpG/Al(OH)3 (N=32) | Month-0, Month-2 Cohort: Placebo (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (FATIGUE) (General disorders) | 7 | 6 | 9 | 9 | 6 | 4 | 14 | 6 | 12 | 13
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (REDNESS) (General disorders) | 2 | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 5 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 10 | 10 | 1 | 9 | 7 | 5 | 6 | 3 | 12 | 4
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (SWELLING) (General disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 4 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (FEVER) (General disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Vaccination site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 4 | 2 | 5 | 2 | 1 | 3 | 2 | 4 | 2 | 4
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (NAUSEA) (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 3 | 0 | 2 | 3 | 1 | 4
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Giardiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5 | 2 | 0 | 2 | 3 | 4 | 4 | 7
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 4 | 5 | 5 | 6 | 6 | 6 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Headache (HEADACHE) (Nervous system disorders) | 6 | 3 | 1 | 6 | 2 | 5 | 12 | 2 | 5 | 9
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study follow up of the Month-0, Month-2 cohort was terminated early due to sponsor decision, with all participants followed up through 6 months after Vaccination 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03572062/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT03572062/SAP_001.pdf